CLINICAL TRIAL: NCT03435146
Title: Safety, Tolerability, and Drug-drug Interactions of Short-course Treatment of Latent Tuberculosis Infection With High-dose Rifapentine and Isoniazid or Standard Isoniazid Preventative Therapy Among HIV-infected Patients Taking Dolutegravir-based Antiretroviral Treatment
Brief Title: Safety Tolerability DDI Short Course Treatment of LTBI Infection With High-dose Rifapentine and Isoniazid or Standard Isoniazid Preventive Therapy in HIV+ Patients (DOLPHIN & DOLPHIN TOO)
Acronym: IMPAACT4TB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Johns Hopkins University (Other); University of California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3HP DTG AUR1-6-212 IMPAACT4TB
Record Dates: First submitted 2017-08-21; First posted 2018-02-15 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Tract Infections; HIV Infections
Keywords: 3HP; LTBI; IMPAACT4TB; DDI; Pharmacokinetics; Dolutegravir
MeSH Terms: conditions — Respiratory Tract Infections; HIV Infections

STUDY DESIGN:
Intervention Model Description: Group 1A:12 ppts will take DTG 50mg/TDF/FTC once daily + once weekly HP for 12 weeks. Semi-intensive PK for DTG,RPT,INH will be collected per protocol.An interim PK, safety,and HIV VL assessment will be performed to ensure that DTG 50mg once daily is safe and meets PK targets.Group 1B:18 ppts will receive either DTG 50mg or dose adjusted DTG + once weekly HP. Semi-intensive PK for DTG,RPT,INH will be collected per protocol.Group 2: 30 ppts will receive DTG at the same dose and frequency as Group 1B. Sparse PK for DTG, safety labs and HIV VL will be measured per protocol.Group 3: 25 ppts who are HIV tx naive will start DTG 50mg/TDF/3TC daily as a FDC tablet + standard of care isoniazid preventive therapy. ART and IPT will start together. Sparse PK for DTG will be collected per protocol.Group 4: 50 ppts who are HIV treatment naive will start DTG 50mg/TDF/3TC daily as a FDC tablet + weekly HP for 12 weeks. ART and 3HP will start together. Sparse PK for DTG will be collected per protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Groups 1,2,3 and 4 (Experimental): Group 1: The first 12 participants (Group 1A) will undergo semi-intensive PK sampling and will be key to determining whether an increased dosing of dolutegravir is required in groups 1B. Group 1B will receive dolutegravir at the new dose (if applicable) and will also undergo semi-intensive PK sampling. All will undergo safety and HIV VL assessments.
  3HP plus DTG +2NRTIs
  Group 2: The next 30 (Group 2) will receive dolutegravir at the new dose and will only have sparse PK sampling. All will undergo safety and HIV VL assessments.
  3HP plus DTG +2NRTIs
  Group 3: The next 25 (Group 3) will receive dolutegravir at the same dose as Group 2 and will only have sparse PK sampling. All will undergo safety and HIV VL assessments.
  IPT plus DTG +2NRTIs
  Group 4: The next 50 (Group 4) will receive dolutegravir at the same dose as Group 2 and will only have sparse PK sampling. All will undergo safety and HIV VL assessments.
  3HP plus DTG +2NRTIs
  Interventions: Combination Product: 3HP plus DTG +2NRTIs

INTERVENTIONS:
Combination Product: 3HP plus DTG +2NRTIs — * HIV treatment: DTG will be dosed as described above and will be given with daily TDF/FTC (Groups 1 and 2) or with TDF/3TC (Groups 3 and 4).
  * LTBI treatment: 3HP will be given once-weekly for a total of 12 doses, with doses as follows:
  Rifapentine: 900 mg; Isoniazid: 900 mg (Groups 1,2 and 4) Isoniazid at standard of care dosing (Group 3)

SUMMARY:
Single-arm, single-center, Phase I/II clinical trial, in four groups. Individuals with HIV infection taking Efavirenz (EFV) and two nucleoside reverse transcriptase inhibitors (NRTI) who have undetectable (Groups 1 and 2) or detectable (Group 3 and 4) HIV viral load and an indication for TPT, will be switched to DTG with tenofovir/emtricitabine (Groups 1 and 2) or lamivudine/tenofovir (Groups 3 and 4). Group 1 and 2 will receive weekly HP for 12 total doses starting 8 weeks after initiating DTG. Individuals who are on an existing DTG-based plus two NRTI ART regimen for at least eight weeks (and have not received efavirenz or nevirapine for at least two months) who have an undetectable HIV viral load may also participate. Individuals with HIV infection who are ART treatment naïve at any HIV viral load level and have an indication for TPT will start DTG and be enrolled to receive standard IPT (Group 3) or HP (Group 4) initiated at the same time as DTG. Group 3 and 4 will be enrolled after follow up of Group 1 and 2 has been completed.

DETAILED DESCRIPTION:
Group 1 (n=30): The first 12 participants (Group 1A) will take dolutegravir 50 milligrams (mg) once daily (with tenofovir/emtricitabine) from Days 1-57. Semi-intensive PK sampling for dolutegravir will be performed on Day 57. Participants will continue once-daily dolutegravir and will receive once-weekly HP for 12 total doses beginning on Day 58. Semi-intensive PK sampling for dolutegravir will be performed on Day 72 (with the 3rd dose of HP) and Day 108 (following the 8th dose of HP). Trough concentrations (CT) will be measured on Days 59, 74, and 78. PK assessments will be performed at weeks 9 and 11 for rifapentine and at week 11 for isoniazid. VL will be measured at baseline and weeks 11 and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E) and creatinine and liver function tests (LFT)) will be obtained at baseline, and weeks 9, 11, 13, 16, 20 and 24.

After the 12 Group 1A participants have completed the second semi-intensive PK visit, an interim PK, safety, and VL assessment will be performed to ensure that the 50 mg once daily dose is safe and meets PK targets. The subsequent 18 participants in Group 1 (Group 1B) will receive either dolutegravir 50 mg or a higher dose of dolutegravir, if dose adjustment is required (e.g. dolutegravir 50 mg twice daily just on HP dosing days, dolutegravir 50 mg twice daily seven days a week, etc.) A second interim evaluation focused on PK will occur after all Group 1B participants have completed the Week 11 semi-intensive PK visit. This evaluation will include all PK data from Group 1A, who will have completed their Week 16 semi-intensive PK visit plus PK data from Group 1B up to and including the Week 11 semi-intensive PK visit.

A third interim evaluation focused on safety and virologic response will occur after all participants (Groups 1A, 1B, and 2) have completed the Week 11 visit. This evaluation will include all safety data and HIV viral load information collected up until that point from all participants.

Group 2 (n=30): These participants will receive dolutegravir and HP at the same doses and dose schedule as the participants in Group 1B. They will undergo safety assessments at baseline and weeks 9, 11, 13, 16, 20 and 24; HIV VL assessments will be performed at baseline and weeks 11 and 24. Sparse (trough) PK samples for dolutegravir will be collected on two occasions.

Group 3 (n=25): The next 25 participants who are ART treatment naïve will start dolutegravir 50 milligrams (mg) once daily (with tenofovir/lamivudine on study Day 0. Sparse PK sampling for trough concentrations (CT) of dolutegravir will be performed on Day 1 (24 hours after taking the first dose of DTG, and before taking the first dose of standard isoniazid). Sparse PK sampling for trough concentrations (CT) of dolutegravir will be performed on Day 24 (Week 3), to parallel 721 hours after the 3rd dose of HP. The final sparse PK sampling for trough concentrations (CT) of dolutegravir will be performed on Day 59 (Week 8), to parallel 721 hours after the 8th dose of HP. HIV VL will be measured at screening, and Weeks 3, 8, 12, 16, and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E) and creatinine and liver function tests (LFT)) will be obtained at baseline. Creatinine will be repeated at Weeks 2, 4, 8, 12, 16 and 24 and LFTs will be repeated at weeks 4, 8, and 12.

Group 4 (n=50): After Group 3 is fully enrolled, another group of 50 participants who are ART treatment naïve will start dolutegravir 50 milligrams (mg) once daily (with tenofovir/lamivudine) on Day 0. They will begin TPT with once weekly HP the day after starting DTG, on Day 1. Sparse PK sampling for trough concentrations (CT) dolutegravir will be performed on Day 1 (24 hours after the first dose of DTG, before the first dose of HP). Sparse PK sampling for trough concentrations (CT) of dolutegravir will be performed on Day 24 (721 hours after the third dose of HP). Sparse PK sampling for trough concentrations (CT) of dolutegravir will be performed on Day 59 (721 hours after the eighth dose of HP). HIV VL will be measured at screening, and Weeks 3, 8, 12, 16, and 24. Safety labs (complete blood count (CBC), urea and electrolytes (U&E) and creatinine and liver function tests (LFT)) will be obtained at baseline. Creatinine will be repeated at Weeks 2, 4, 8, 12, 16, and 24, and LFTs will be repeated at weeks 4, 8, and 12.

1 (+/- 24 hours)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Weight > 50 kg
3. Documented HIV infection*
4. At least 8 weeks of HIV treatment with efavirenz or dolutegravir plus two NRTI, or ART treatment naïve, depending upon the enrolling treatment Group
5. Undetectable or detectable HIV-1 viral load, depending upon the enrolling treatment Group

Exclusion Criteria:

1. Confirmed or suspected TB disease
2. Likely to move from the study area during the study period
3. Known exposure to TB cases with known or suspected resistance to isoniazid or rifampicin in the source case
4. TB treatment within the past year
5. TB preventive therapy within the last year
6. Sensitivity or intolerance to isoniazid or rifamycins
7. On nevirapine, etravirine, rilpivirine, PI-based, or raltegravir-containing ART regimens
8. Suspected acute hepatitis or known chronic liver disease; severe hepatic impairment (Class C or greater) as determined by Child Pugh classification
9. ALT≥ 3 times the upper limit of normal (ULN)
10. Total bilirubin ≥ 2.5 times the ULN
11. Absolute neutrophil count (ANC) ≤ 750 cells/mm3
12. Creatinine clearance < 50 ml/min
13. Pregnancy or breastfeeding
14. Women of childbearing potential who are unable or unwilling to use contraception
15. Self-reported alcohol use exceeding 28 units per week for men, or 21 units for women
16. Karnofsky status < 80
17. On prohibited medications e.g. dofetilide (see Appendix 1)
18. Known porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
PK sampling of Dolutegravir - Ctau | PK sampling at Week 9 (Group 1), Week 11 (Groups 1 and 2) and Week 16 (Groups 1 and 2); Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Trough concentration in the presence or absence of once weekly HP
PK sampling of Dolutegravir - AUC parameter | PK sampling at Week 9 (Group 1), Week 11 (Groups 1 and 2) and Week 16 (Groups 1 and 2); Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Daily area under curve (AUC) in the presence or absence of once weekly HP
PK sampling of Dolutegravir - Cmin parameter | PK sampling at Week 9 (Group 1), Week 11 (Groups 1 and 2) and Week 16 (Groups 1 and 2); Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Minimum concentration (Cmin) in the presence or absence of once weekly HP
Adverse Events (Primary) | Adverse events to be collected from Week 1 through Week 24, to be reported throughout the trial
  Grade 3 or higher adverse events (AE)

SECONDARY OUTCOMES:
HIV-1 RNA viral load | HIV viral load to be measured in Groups 1 and 2 at screening, weeks 11 and 24; and in Groups 3 and 4 at screening and weeks 3, 8, 12 and 24, to be reported at end of trial
  HIV-1 RNA viral load (copies/ml)
PK sampling of RPT - AUC parameter | PK sampling at Weeks 9 and 11 (Group 1); and Week 11 (Group 2), Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Area under curve (AUC).
PK sampling of RPT - Cmax parameter | PK sampling at Weeks 9 and 11 (Group 1); and Week 11 (Group 2), Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Maximum concentration (Cmax).
PK sampling of RPT - Cmin parameter | PK sampling at Weeks 9 and 11 (Group 1); and Week 11 (Group 2), Day 1 (Groups 3 and 4), Week 3 (Groups 3 and 4) and Week 8 (Groups 3 and 4) to be reported at end of trial
  Minimum concentration (Cmax).
PK sampling of INH - AUC parameter | PK sampling at Week 11(Group 1 only), to be reported at end of trial
  Area under curve (AUC). NAT 2 acetylator status to be taken into account
PK sampling of INH - Cmax parameter | PK sampling at Week 11(Group 1 only), to be reported at end of trial
  Maximum concentration (Cmax). NAT 2 acetylator status to be taken into account
PK sampling of INH - Cmin parameter | PK sampling at Week 11(Group 1 only), to be reported at end of trial
  Minimum concentration (Cmin). NAT 2 acetylator status to be taken into account
DTG Dose selection | Post Group 1A. Dose will be selected once Group 1a participants' PK data have been analyzed. The dolutegravir dose may be adjusted according to PK results. If warranted, the revised dose will be administered to Groups 1B and 2.
  Dose options for DTG with once-weekly HP derived by simulation using nonlinear mixed effects models.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Churchyard, MBBCh PhD, Principal Investigator — Global CEO: The Aurum Institute, NPC
Locations (1):
- The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
To be shared amongst the collaborators on shared database when study starts and is complete.
  Results will be disseminated via conferences and publication by scientific peer reviewed journal(s)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Pre-study start: Study protocol and Informed Consent Form to collaborators on SharePoint).
  Post-study completion: Clinical Study Report, Results with Statistical Analysis will be shared with scientific peer reviewed journal(s) and collaborators.
Access Criteria: Password protected and user defined credentials (Pre-study via SharePoint)
  Open access (Post-study completion)

REFERENCES:
- [Derived] Weld ED, Beattie T, Moodley J, Mapendere M, Salles I, Solans BP, Nonyane BAS, Wiesner L, Nielson T, Edward VA, Chihota V, Savic RM, Dooley KE, Chaisson RE, Churchyard GJ; DOLPHIN-TOO Study Team; Unitaid IMPAACT4TB Research Group. Simultaneous initiation of dolutegravir-based antiretroviral therapy and once-weekly rifapentine and isoniazid for tuberculosis prevention in antiretroviral-naive people with HIV: an open-label, non-randomised, phase 1/2 trial. Lancet HIV. 2025 Jun;12(6):e428-e439. doi: 10.1016/S2352-3018(25)00002-5. Epub 2025 May 8. PMID 40349709
- [Derived] Jarrett RT, van der Heijden Y, Shotwell MS, Chihota V, Marzinke MA, Chaisson RE, Dooley KE, Churchyard GJ. High Isoniazid Exposures When Administered with Rifapentine Once Weekly for Latent Tuberculosis in Individuals with Human Immunodeficiency Virus. Antimicrob Agents Chemother. 2023 Feb 16;67(2):e0129722. doi: 10.1128/aac.01297-22. Epub 2023 Jan 9. PMID 36622148
- [Derived] Dooley KE, Savic R, Gupte A, Marzinke MA, Zhang N, Edward VA, Wolf L, Sebe M, Likoti M, Fyvie MJ, Shibambo I, Beattie T, Chaisson RE, Churchyard GJ; DOLPHIN Study Team. Once-weekly rifapentine and isoniazid for tuberculosis prevention in patients with HIV taking dolutegravir-based antiretroviral therapy: a phase 1/2 trial. Lancet HIV. 2020 Jun;7(6):e401-e409. doi: 10.1016/S2352-3018(20)30032-1. Epub 2020 Mar 30. PMID 32240629

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03435146/Prot_SAP_000.pdf